CLINICAL TRIAL: NCT05448066
Title: Molecular Allergen Based Diagnosis Impact on Clinical Efficacy of Aeroallergen Immunotherapy- a Pragmatic Randomized Clinical Trial
Brief Title: Molecular Allergen Component Resolved Diagnosis to Decide Immunotherapy
Acronym: CRD-AIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Sociedade Portuguesa de Alergologia e Imunologia Clinica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2017-21
Record Dates: First submitted 2022-04-21; First posted 2022-07-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-06

CONDITIONS: Asthma; Rhinitis, Allergic
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard diagnosis (Active Comparator): Patients followed in the allergy clinic with indication for allergen immunotherapy using only standard diagnosis.
  Interventions: Diagnostic Test: Standard diagnosis
- CRD diagnosis (Experimental): Patients followed in the allergy clinic with indication for allergen immunotherapy decided with standard diagnostic tools and molecular based diagnosis.
  Interventions: Diagnostic Test: Component resolved diagnosis

INTERVENTIONS:
Diagnostic Test: Component resolved diagnosis — Physicians in this group will have access to allergen molecular component sensitization profile, using ImmunoCAP ISAC E112i and to all standard diagnostic tolls
  Arms: CRD diagnosis
Diagnostic Test: Standard diagnosis — Physicians will only have access to standard diagnostic tools namely skin prick tests and sIgE sensitization (not molecular IgE) and clinical history.
  Arms: Standard diagnosis

SUMMARY:
Allergen immunotherapy (AIT) is used for the control of allergic diseases that are not completely responsive to avoidance strategies and/or pharmacotherapy. It is also considered the main treatment with the potential to modify allergic disease evolution. It's efficacy and safety in allergic rhinitis and asthma is supported by large systematic reviews and is recommended as a cornerstone treatment option in allergic disease. Molecular based allergy diagnosis has greatly evolved and the knowledge of molecular allergen sensitization pattern has been used to better define the allergen extract composition of AIT. However, uncertainty remains if this strategy is related to an increase of efficacy. Regulation of allergen extracts for allergen immunotherapy are currently underway in Europe, but there is still lack of standardization of relevant allergens and important differences are seen between allergenic contents.

Therefore, we aim to evaluate, in a real-life setting, the impact of using molecular-based diagnosis versus standard diagnostic tools in the efficacy of aeroallergen immunotherapy, using a pragmatic randomized controlled trial design and also to address the impact of the discrepancy between individual aeroallergen sensitization profiles and the major allergen molecular content of aeroallergen immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with medical indication for aeroallergen immunotherapy(AIT) for allergic rhinoconjunctivitis or asthma, accordingly to the AIT guidelines;
* Over 5 years of age;
* Evidence of IgE-sensitization (positive skin prick tests and / or serum specific-IgE)
* Patients have indication to AIT to house dust mites and/or grass pollen, association with other allergens is not an exclusion criteria

Exclusion Criteria:

* Previously performed allergen immunotherapy
* Need the use of molecular allergen diagnosis to decide treatment and diagnostic strategy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of combined symptom and medication score (CSMS) at 52 weeks | 0 to 52 weeks
  Differences, in the mean change at 52 weeks, of CSMS between groups that were treated with AIT in the component resolved diagnosis versus standard diagnosis groups. CSMS is the sum of the daily symptom score (dSS, score 0 to 3) plus daily medication score (dMS; score 0 to 6)
Change of combined symptom and medication score (CSMS) at 24 weeks | 0 to 24 weeks
  Difference, in the mean change at 24 weeks, of CSMS between groups were treated with AIT in the component resolved diagnosis versus standard diagnosis groups.
Change of rhinitis symptoms using visual analogue scale at 52 weeks | 0 to 52 weeks
  Difference between groups(control vs intervention) in the mean change at 52 weeks, in the psychometric response scale. This scale is used to assess rhinoconjunctivitis discomfort and its impacts on symptom severity and need of treatment.
Change of rhinitis symptoms using visual analogue scale at 24 weeks | 0 to 24 weeks
  Difference between groups(control vs intervention) in the mean change at 52 weeks, in the psychometric response scale. This scale is used to assess rhinoconjunctivitis discomfort and its impacts on symptom severity and need of treatment.

SECONDARY OUTCOMES:
Change in Control of Allergic Rhinitis and Asthma Test (CARAT) at 52 weeks | 0 to 52 weeks
  Differences between groups (control vs intervention) in the mean change at 52 weeks in the scores obtained on the self-administered Portuguese validated questionnaire that assess symptoms and control of both allergic rhinitis and asthma in the previous 4 weeks. The final score ranges from 0 to 30, with scores over 24 indicating good control of asthma and allergic rhinitis, a four-point changes will be considered the minimal important difference
Change in Control of Allergic Rhinitis and Asthma Test (CARAT) at 24 weeks | 0 to 24 weeks
  Differences between groups (control vs intervention) in the mean change at 24 weeks in the scores obtained on the self-administered Portuguese validated questionnaire that assess symptoms and control of both allergic rhinitis and asthma in the previous 4 weeks. The final score ranges from 0 to 30, with scores over 24 indicating good control of asthma and allergic rhinitis, a four-point changes will be considered the minimal important difference.
Change in Asthma Control Test (ACT) at 52 weeks | 0 to 52 weeks
  Differences between control and intervention group of change in the self-report questionnaire regarding asthma symtoms that includes 5 items assessing each of the following for the previous 4 weeks. ACT score ranges from 5 (poor control of asthma) to 25 (complete control of asthma)
Change in Asthma Control Test (ACT) at 24 weeks | 0 to 24 weeks
  Differences between control and intervention group of change in the self-report questionnaire regarding asthma symtoms that includes 5 items assessing each of the following for the previous 4 weeks. ACT score ranges from 5 (poor control of asthma) to 25 (complete control of asthma)
Change in quality of life related with rhinitis and asthma at 52 weeks | 0 to 52 weeks
  Difference between groups regarding self-administered version of Rhinoconjunctivitis Quality of Life Questionnaire which is validated in Portuguese for patients over 12 years at 52 weeks. A change greater than 0.5 will be considered a critically clinically significant difference
Change in quality of life related with rhinitis and asthma at 24 weeks | 0 to 24 weeks
  Differences between groups regarding the self-administered version of Rhinoconjunctivitis Quality of Life Questionnaire which is validated in Portuguese for patients over 12 years at 24 weeks. A change greater than 0.5 will be considered a critically clinically significant difference
Change in ESPIA score- patient reported opinion allergen immunotherapy at 52 weeks | 0 to 52 weeks
  Differences between intervention and control groups in the self-administered questionnaire with 16 questions distributed in 4 dimensions: perception of effectiveness, activities and environment, cost-benefit balance and general satisfaction at 52 weeks
Change in ESPIA score- patient reported opinion allergen immunotherapy at 24 weeks | 0 to 24 weeks
  Differences in the self-administered questionnaire with 16 questions distributed in 4 dimensions: perception of effectiveness, activities and environment, cost-benefit balance and general satisfaction at 24 weeks
Change in the cost impact between groups | 0 and 52 weeks
  Direct and indirect healthcare related costs will be assessed in each of the groups before and after treatment and compared

CONTACTS AND LOCATIONS:
Overall Officials: Diana Silva, Principal Investigator — Faculty of Medicine Porto University
Locations (1):
- Faculty of Medicine Porto University/Centro Hospitalar de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
All data

REFERENCES:
- [Background] Roberts G, Pfaar O, Akdis CA, Ansotegui IJ, Durham SR, Gerth van Wijk R, Halken S, Larenas-Linnemann D, Pawankar R, Pitsios C, Sheikh A, Worm M, Arasi S, Calderon MA, Cingi C, Dhami S, Fauquert JL, Hamelmann E, Hellings P, Jacobsen L, Knol EF, Lin SY, Maggina P, Mosges R, Oude Elberink JNG, Pajno GB, Pastorello EA, Penagos M, Rotiroti G, Schmidt-Weber CB, Timmermans F, Tsilochristou O, Varga EM, Wilkinson JN, Williams A, Zhang L, Agache I, Angier E, Fernandez-Rivas M, Jutel M, Lau S, van Ree R, Ryan D, Sturm GJ, Muraro A. EAACI Guidelines on Allergen Immunotherapy: Allergic rhinoconjunctivitis. Allergy. 2018 Apr;73(4):765-798. doi: 10.1111/all.13317. Epub 2017 Oct 30. PMID 28940458
- [Background] Matricardi PM, Dramburg S, Potapova E, Skevaki C, Renz H. Molecular diagnosis for allergen immunotherapy. J Allergy Clin Immunol. 2019 Mar;143(3):831-843. doi: 10.1016/j.jaci.2018.12.1021. PMID 30850070
- [Background] Dhami S, Nurmatov U, Arasi S, Khan T, Asaria M, Zaman H, Agarwal A, Netuveli G, Roberts G, Pfaar O, Muraro A, Ansotegui IJ, Calderon M, Cingi C, Durham S, van Wijk RG, Halken S, Hamelmann E, Hellings P, Jacobsen L, Knol E, Larenas-Linnemann D, Lin S, Maggina P, Mosges R, Oude Elberink H, Pajno G, Panwankar R, Pastorello E, Penagos M, Pitsios C, Rotiroti G, Timmermans F, Tsilochristou O, Varga EM, Schmidt-Weber C, Wilkinson J, Williams A, Worm M, Zhang L, Sheikh A. Allergen immunotherapy for allergic rhinoconjunctivitis: A systematic review and meta-analysis. Allergy. 2017 Nov;72(11):1597-1631. doi: 10.1111/all.13201. Epub 2017 Jul 14. PMID 28493631